CLINICAL TRIAL: NCT01697410
Title: A Multicenter,Prospective,Randomized,Controlled,Double Blind Study in China to Evaluate the Effect of Terlipressin in Patients With Septic Shock
Brief Title: Continuos Terlipressin Infusion in Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangdong Province, Department of Science and Technology (Other Government); Second Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Chinese PLA General Hospital (Other); Beijing 302 Hospital (Other); Shanghai Changzheng Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Xiangya Hospital of Central South University (Other); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Bengbu Medical University (Other); Guangxi Medical University (Other); Jinling Hospital, China (Other); West China Hospital (Other); Hainan People's Hospital (Other); Xi'an Jiaotong University (Other); China Medical University, China (Other); First People's Hospital of Foshan (Other); ZhuHai Hospital (Other)
Responsible Party: Principal Investigator, Guan XiangDong, director of surgical intensive care unit, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012A080204018;2007015
Record Dates: First submitted 2012-08-28; First posted 2012-10-02 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Terlipressin; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- terlipressin (Experimental)
  Interventions: Drug: Terlipressin
- norepinephrine (Active Comparator)
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Terlipressin — continuous infusion of terlipressin (0.66ug/min-2.66ug/min) ,dosage modified acorrding to blood pressure
  Arms: terlipressin
Drug: Norepinephrine — continuous infusion with dose 7.5ug/min-30ug/min,modified acorrding to blood pressure
  Arms: norepinephrine

SUMMARY:
The purpose of this study is to evaluate the efficacy of terlipressin for treating septic shock.

DETAILED DESCRIPTION:
Septic shock is the most common cause of death in intensive care units and has a mortality rate of 40 to 60%.Vasopressin is commonly used as an adjunct to catecholamines to support blood pressure in refractory septic shock.Recently small sample clinical study suggest that Terlipressin,a vasopressin analogues, was effective in reversing sepsis-induced arterial hypotension and in reducing norepinephrine requirements.But its effect on mortality is unknown.Invesgators hypothesized that Terlipressin as compared with norepinephrine would decrease mortality among patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock was defined by the presence of two or more diagnostic criteria for the systemic inflammatory responsesyndrome, proven or suspected infection, and hypotension (exclusion of hypertention other than sepsis)

Exclusion Criteria:

* organ transplantation;
* pregancy or breast-feeding;
* malignancy or other irreversible disease or condition for which has a poor prognosis;
* acute coronary syndrome;
* chronic heart failure(NYHA III or IV)/cardiogenic shock;
* acute mesenteric ischemia;
* greater than 48 hours had elapsed since the patient met entry criteria;
* estimation of incomplite treament due to financial problem;
* use of terlipressin for blood pressure support before entry;
* Raynaud's phenomenon, systemic sclerosis or vasospastic diathesis;
* registration of other clinical trial which will affect the outcome of the current study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
28-day Mortality | 28-days
  The prospectively defined primary end point was death from any cause and was assessed 28 days after the start of the infusion

SECONDARY OUTCOMES:
SOFA score | 7 days
  SOFA score was measured on day0-7 after the start of the infusion in both groups
days alive and free of vasopressor | during the first 28 days after the start of the infusion
  Days of vasopressor were recorded after the start of the infusion in both groups.
90-day mortality | 90 days after the start of the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Guan XiangDong, doctor, Study Chair — first affiliated hospital SunYetSen university; liu ZiMeng, M.D, Study Director — first affiliated hospital ,SunYetSen university; Si Xiang, M.D., Principal Investigator — first affiliated hospital ,SunYetSen university; Chen Juan, M.D., Principal Investigator — first affiliated hospital ,SunYetSen university
Locations (1):
- Surgical intensive care unit, 1st affiliated hospital of Sun Yat-sen university, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu ZM, Chen J, Kou Q, Lin Q, Huang X, Tang Z, Kang Y, Li K, Zhou L, Song Q, Sun T, Zhao L, Wang X, He X, Wang C, Wu B, Lin J, Yuan S, Gu Q, Qian K, Shi X, Feng Y, Lin A, He X; Study Group of investigators; Guan XD. Terlipressin versus norepinephrine as infusion in patients with septic shock: a multicentre, randomised, double-blinded trial. Intensive Care Med. 2018 Nov;44(11):1816-1825. doi: 10.1007/s00134-018-5267-9. Epub 2018 Jul 3. PMID 29971593